CLINICAL TRIAL: NCT03114254
Title: A Phase II Trial of Cabazitaxel Chemotherapy in Relapsed Locally Advanced &/or Metastatic Carcinoma of the Penis
Brief Title: A Trial of Cabazitaxel Chemotherapy in Relapsed Locally Advanced &/or Metastatic Carcinoma of the Penis
Acronym: JAVA-P
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ON/2012/4233; 2014-002336-14 (EudraCT Number); CabazL05881 (Other Grant/Funding Number: Sanofi)
Record Dates: First submitted 2014-10-30; First posted 2017-04-14 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Penile Neoplasm
Keywords: Recurrent; Locally advanced; Metastatic
MeSH Terms: conditions — Penile Neoplasms; Recurrence; Neoplasm Metastasis | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel (Experimental): Six cycles of chemotherapy comprising:
  Cabazitaxel 25mg/m2 to be repeated at intervals of 21 days
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel — Six cycles of chemotherapy comprising:
  Cabazitaxel 25mg/m2 to be repeated at intervals of 21 days.
  Other Names: Jetvana

SUMMARY:
An evaluation of the activity of cabazitaxel chemotherapy in relapsed cancer of the penis. Safety and tolerability will be monitored and survival will be assessed. It is hypothesised that cabazitaxel is useful in increasing progression free survival in relapsed penile cancer.

DETAILED DESCRIPTION:
First line treatment of penile cancer often combines Docetaxel, Cisplatin and 5Fluouracil (5FU) and there is currently no United Kingdom standard second line agent. Carbazitaxel has been shown to kill both taxane resistant and sensitive cells. JAVA-P is a phase two, single arm study of the use of carbazitaxel for relapsed, locally advanced or metastatic carcinoma of the penis. Seventeen patients will be recruited over two years, with adverse events and progression free survival being assessed. Results may indicate the need for larger studies to evaluate carbazitaxel as a first line agent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven squamous cell carcinoma of the penis
* Performance status ECOG 0-2
* Written informed consent
* Measurable disease as per RECIST 1.1
* Fit to receive cabazitaxel as second line chemotherapy
* Previously received TPF or cisplatin-5FU as first line systemic chemotherapy for penile cancer
* Adequate organ function as evidenced by the following peripheral blood counts and serum biochemistry at enrollment:

  * Neutrophils ≥1.5 x 109/L
  * Haemoglobin ≥10 g/dL
  * Platelets ≥100 x 109/L
  * Total bilirubin <1.5 upper limit of normal (ULN)
  * Alanine aminotransferase/serum glutamate pyruvate transaminase (ALT/SGPT) ≤1.5 x ULN
  * Serum creatinine ≤1.5 x ULN. (If creatinine is 1.0-1.5 x ULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with a creatinine clearance <60 ml/min should be excluded.)

Exclusion Criteria:

* Pure veruccous carcinoma of the penis
* Squamous carcinoma of the urethra
* T1 N1 M0 disease
* T2 N1 M0 disease
* Unfit for this regimen (as assessed by the multidisciplinary team)
* Contraindication to chemotherapy
* ECOG Performance Status > 2
* Active Grade ≥2 peripheral neuropathy
* Active secondary cancers
* Other concurrent serious illness or medical conditions
* Electrocardiogram (ECG) evidence of uncontrolled cardiac arrhythmias, angina pectoris, and/or hypertension, history of congestive heart failure, or myocardial infarction within last 6 months.
* Uncontrolled diabetes mellitus.
* History of severe hypersensitivity reaction (≥grade 3) to docetaxel
* History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs
* Active infection requiring systemic antibiotic or anti-fungal medication
* Participation in another clinical trial with any investigational drug within 30 days prior to study registration.
* Concurrent or planned treatment with strong inhibitors of cytochrome P450 3A4/5. A 1-week washout period is necessary for patients who are already on these treatments.
* Concurrent or planned treatment with strong inducers of cytochrome P450 3A4/5. A 1-week washout period is necessary for patients who are already on these treatments.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-12-05 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

PRIMARY OUTCOMES:
Complete response | 18 weeks
  Complete response recorded from the start of the treatment to completion of 6 cy-cles of treatment determined by radiological response assessment
Partial response | 18 weeks
  Partial response recorded from the start of the treatment to completion of 6 cy-cles of treatment determined by radiological response assessment

SECONDARY OUTCOMES:
Progression free survival | Until patient progresses, which is approximately 6 weeks after randomisation
  Progression free survival defined as the time from registration to the first of one of the following: development of radiological disease progression (RECIST 1.1) or death from any cause
Overall survival | Until patient dies, which is approximately 3 months after randomisation
  Overall survival defined as time from registration to the date of death due to from any cause
Acute toxicity (Defined by number of CTCAE v4.03 Adverse Events, Adverse Reactions and by grades and the worst grade). | After each cycle (every 3 weeks) for maximally 6 cycles therefore 18 weeks whilst on treatment and at the 3 month visit timepoint
  Acute toxicity (Defined by number of CTCAE v4.03 Adverse Events, Adverse reactions and by grades experienced by the patient collected at study visits and recorded on an Adverse Event Case report form. .
Late toxicity (Defined by number of CTCAE v4.03 Adverse Events, Adverse Reactions and by grades and the worst grade). | From 3 months post treatment Cycle 1 Day 1 to up to 6 months recorded at the 3 month and 6 month timepoint.
  Late toxicity (Defined by number of CTCAE v4.03 Adverse Events, Adverse reactions and by grades experienced by the patient collected at study visits and recorded on an Adverse Event Case report form. .

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bahl, Principal Investigator — University Hospitals Bristol and Weston NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Bristol Haematology and Oncology Centre, Horfield Road, Bristol
  - Universitty College Hospitals NHS Trust, London

REFERENCES:
- [Background] Seixas AL, Ornellas AA, Marota A, Wisnescky A, Campos F, de Moraes JR. Verrucous carcinoma of the penis: retrospective analysis of 32 cases. J Urol. 1994 Nov;152(5 Pt 1):1476-8; discussion 1478-9. doi: 10.1016/s0022-5347(17)32450-3. PMID 7933188
- [Background] Soria JC, Fizazi K, Piron D, Kramar A, Gerbaulet A, Haie-Meder C, Perrin JL, Court B, Wibault P, Theodore C. Squamous cell carcinoma of the penis: multivariate analysis of prognostic factors and natural history in monocentric study with a conservative policy. Ann Oncol. 1997 Nov;8(11):1089-98. doi: 10.1023/a:1008248319036. PMID 9426328
- [Background] Cubilla AL, Ayala MT, Barreto JE, Bellasai JG, Noel JC. Surface adenosquamous carcinoma of the penis. A report of three cases. Am J Surg Pathol. 1996 Feb;20(2):156-60. doi: 10.1097/00000478-199602000-00003. PMID 8554104
- [Background] Somogyi L, Kalman E. Metaplastic carcinoma of the penis. J Urol. 1998 Dec;160(6 Pt 1):2152-3. doi: 10.1097/00005392-199812010-00059. No abstract available. PMID 9817349
- [Background] Tomic S, Warner TF, Messing E, Wilding G. Penile Merkel cell carcinoma. Urology. 1995 Jun;45(6):1062-5. doi: 10.1016/s0090-4295(99)80134-4. PMID 7771012
- [Background] Kim ED, Kroft S, Dalton DP. Basal cell carcinoma of the penis: case report and review of the literature. J Urol. 1994 Nov;152(5 Pt 1):1557-9. doi: 10.1016/s0022-5347(17)32471-0. PMID 7933201
- [Background] Bundrick WS, Culkin DJ, Mata JA, Gonzalez E, Zitman R, Venable DD. Penile malignant melanoma in association with squamous cell carcinoma of the penis. J Urol. 1991 Nov;146(5):1364-5. doi: 10.1016/s0022-5347(17)38096-5. PMID 1942294
- [Background] Oppenheim AR. Sebaceous carcinoma of the penis. Arch Dermatol. 1981 May;117(5):306-7. No abstract available. PMID 7224661
- [Background] Wood EW, Gardner WA Jr, Brown FM. Spindle cell squamous carcinoma of the penis. J Urol. 1972 Jun;107(6):990-1. doi: 10.1016/s0022-5347(17)61190-x. No abstract available. PMID 5033986
- [Background] Srinivas V, Morse MJ, Herr HW, Sogani PC, Whitmore WF Jr. Penile cancer: relation of extent of nodal metastasis to survival. J Urol. 1987 May;137(5):880-2. doi: 10.1016/s0022-5347(17)44281-9. PMID 3573181
- [Background] Ravi R. Correlation between the extent of nodal involvement and survival following groin dissection for carcinoma of the penis. Br J Urol. 1993 Nov;72(5 Pt 2):817-9. doi: 10.1111/j.1464-410x.1993.tb16273.x. PMID 8281416
- [Background] Slaton JW, Morgenstern N, Levy DA, Santos MW Jr, Tamboli P, Ro JY, Ayala AG, Pettaway CA. Tumor stage, vascular invasion and the percentage of poorly differentiated cancer: independent prognosticators for inguinal lymph node metastasis in penile squamous cancer. J Urol. 2001 Apr;165(4):1138-42. PMID 11257655
- [Background] Solsona E, Iborra I, Rubio J, Casanova JL, Ricos JV, Calabuig C. Prospective validation of the association of local tumor stage and grade as a predictive factor for occult lymph node micrometastasis in patients with penile carcinoma and clinically negative inguinal lymph nodes. J Urol. 2001 May;165(5):1506-9. PMID 11342906
- [Background] Hussein AM, Benedetto P, Sridhar KS. Chemotherapy with cisplatin and 5-fluorouracil for penile and urethral squamous cell carcinomas. Cancer. 1990 Feb 1;65(3):433-8. doi: 10.1002/1097-0142(19900201)65:33.0.co;2-g. PMID 2297633
- [Background] Shammas FV, Ous S, Fossa SD. Cisplatin and 5-fluorouracil in advanced cancer of the penis. J Urol. 1992 Mar;147(3):630-2. doi: 10.1016/s0022-5347(17)37327-5. PMID 1538445
- [Background] Ahmed T, Sklaroff R, Yagoda A. Sequential trials of methotrexate, cisplatin and bleomycin for penile cancer. J Urol. 1984 Sep;132(3):465-8. doi: 10.1016/s0022-5347(17)49693-5. PMID 6206239
- [Background] Gagliano RG, Blumenstein BA, Crawford ED, Stephens RL, Coltman CA Jr, Costanzi JJ. cis-Diamminedichloroplatinum in the treatment of advanced epidermoid carcinoma of the penis: a Southwest Oncology Group Study. J Urol. 1989 Jan;141(1):66-7. doi: 10.1016/s0022-5347(17)40590-8. PMID 2642312
- [Background] Sklaroff RB, Yagoda A. Cis-diamminedichloride platinum II (DDP) in the treatment of penile carcinoma. Cancer. 1979 Nov;44(5):1563-5. doi: 10.1002/1097-0142(197911)44:53.0.co;2-s. PMID 498030
- [Background] Theodore C, Skoneczna I, Bodrogi I, Leahy M, Kerst JM, Collette L, Ven K, Marreaud S, Oliver RDT; EORTC Genito-Urinary Tract Cancer Group. A phase II multicentre study of irinotecan (CPT 11) in combination with cisplatin (CDDP) in metastatic or locally advanced penile carcinoma (EORTC PROTOCOL 30992). Ann Oncol. 2008 Jul;19(7):1304-1307. doi: 10.1093/annonc/mdn149. Epub 2008 Apr 15. PMID 18417462
- [Background] Oudard S. TROPIC: Phase III trial of cabazitaxel for the treatment of metastatic castration-resistant prostate cancer. Future Oncol. 2011 Apr;7(4):497-506. doi: 10.2217/fon.11.23. PMID 21463139